CLINICAL TRIAL: NCT06701136
Title: A Clinical Study to Evaluate the Drug-Drug Interaction and Food Effect of Sudapyridine(WX-081) Tablet With Itraconazole and Rifampin in Healthy Chinese Adult Volunteers
Brief Title: Drug-Drug Interaction and Food Effect of Sudapyridine(WX-081) With Itraconazole and Rifampin in Healthy Chinese Adults
Acronym: WX081-DDI
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Jiatan Pharmatech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JYP0081M103; CTR20221162 (Other: China CDE Clinical Trial Registration Platform)
Record Dates: First submitted 2024-11-18; First posted 2024-11-22 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Rifampicin-Resistant Pulmonary Tuberculosis Patients
MeSH Terms: interventions — sudapyridine; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sudapyridine (WX-081) Alone (Experimental): Participants will receive Sudapyridine (WX-081) tablets orally at a specified dose once daily for 10 days (in Study A and Study B) or once under fasting and fed conditions (in Study C). Pharmacokinetic sampling and safety assessments will be conducted.
  Interventions: Drug: Sudapyridine
- Sudapyridine (WX-081) Combined with Itraconazole or Rifampin (Experimental): Participants will receive Sudapyridine (WX-081) tablets orally at a specified dose once daily for 7 days while co-administered with itraconazole (Study A) or rifampin (Study B). Pharmacokinetic sampling and safety assessments will be conducted.
  Interventions: Drug: Sudapyridine; Drug: Itraconazole; Drug: Rifampin

INTERVENTIONS:
Drug: Sudapyridine — In Study A, Cycle 1 (D1-D10): Participants will take Sudapyridine (WX-081) 300 mg once daily after breakfast. Cycle 2 (D11-D14): Participants will take Sudapyridine 300 mg once daily after breakfast with itraconazole 200 mg daily; an additional itraconazole dose (200 mg) will be given after dinner on D11. In Study B, Cycle 1 (D1): Participants will take Sudapyridine 450 mg as a single dose after breakfast. Cycle 2 (D22): Participants will take Sudapyridine 450 mg with rifampin 600 mg daily (D15-D27). In Study C, Cycle 1 (D1): Sudapyridine 450 mg will be given fasting; Cycle 2 (D15): after a high-fat breakfast.
Drug: Itraconazole — In Study A: Participants will receive itraconazole capsules at 200 mg orally once daily after breakfast during Cycle 2 (D11-D14). An additional dose of itraconazole (200 mg) will be administered after dinner on D11.
  Arms: Sudapyridine (WX-081) Combined with Itraconazole or Rifampin
Drug: Rifampin — In Study B: Participants will receive rifampin capsules at 600 mg orally once daily under fasting conditions during Cycle 2 (D15-D27).
  Arms: Sudapyridine (WX-081) Combined with Itraconazole or Rifampin

SUMMARY:
The goal of this clinical trial is to learn how Sudapyridine (WX-081) tablets interact with other drugs and how food intake affects its pharmacokinetics in healthy Chinese adults. The main questions it aims to answer are:

How does itraconazole (a strong CYP3A inhibitor) affect the pharmacokinetics of Sudapyridine? How does rifampin (a strong CYP3A inducer) affect the pharmacokinetics of Sudapyridine? How does food intake influence the pharmacokinetics of Sudapyridine?

Participants will:

Take Sudapyridine alone, with itraconazole, with rifampin, and under fed and fasting conditions based on a predefined sequence.

Attend multiple clinic visits for blood sample collection and safety evaluations.

Researchers will compare the pharmacokinetic parameters of Sudapyridine under these conditions to determine the impact of drug-drug interactions and food.

DETAILED DESCRIPTION:
This open-label, single-center, interventional clinical study aims to assess the pharmacokinetics, safety, and tolerability of Sudapyridine (WX-081) tablets when administered with itraconazole, rifampin, and under fed and fasting conditions in healthy Chinese adults.

The primary objectives are:

To evaluate the effects of itraconazole, a potent CYP3A inhibitor, on the pharmacokinetics of Sudapyridine.

To assess the impact of rifampin, a strong CYP3A inducer, on the pharmacokinetics of Sudapyridine.

To investigate the influence of food on the pharmacokinetics of Sudapyridine. The study will adopt a crossover design with participants assigned to various treatment sequences to ensure comprehensive evaluation of the drug-drug interactions and food effects. The secondary objectives include determining safety profiles and providing key insights for dose adjustments and clinical use of Sudapyridine in subsequent trials.

The results from this trial will contribute to understanding the pharmacokinetic and safety characteristics of Sudapyridine, supporting its further clinical development.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy male or female adults of Chinese nationality, aged 18-50 years (including 18 and 50).

Male participants must weigh at least 50 kg, and female participants at least 45 kg. Body mass index (BMI) should be between 18 and 28 kg/m² (including 18 and 28), and weight (kg)/height (m²).

Participants must undergo a comprehensive physical examination, 12-lead ECG, vital signs assessment, and laboratory tests. Results must be normal or deemed clinically insignificant by the investigator, meeting the following:

12-lead ECG must show QTcF ≤ 450 ms (≤ 200 ms for A Study), QRS duration ≤ 120 ms, and PR interval ≤ 200 ms. PR elongation may allow entry if deemed clinically insignificant by the investigator.

Participants (including their partners) must agree to use effective contraception from the date of screening to 6 months after the last study drug administration and must avoid sperm/egg donation during this period.

Exclusion Criteria:

* Participants with central nervous system, cardiovascular, gastrointestinal, urinary, respiratory, musculoskeletal, endocrine, or hematologic diseases or other chronic/acute diseases, or those with significant surgical history affecting drug absorption, distribution, metabolism, or excretion.

Participants with conditions that increase the risk of QT prolongation, or with a family history of sudden cardiac death (<40 years old) or other hereditary diseases.

Clinically significant laboratory abnormalities at screening, including:

ALT/AST/TBIL values exceeding 2 times the upper limit of normal. Estimated creatinine clearance (ClCr) < 60 mL/min. Participants with urinary system disorders. Use of any prescription or over-the-counter drugs, supplements, or herbal products within 2 weeks before dosing that may affect the study evaluation.

Known allergy to Sudapyridine (WX-081) or other related compounds. Participants positive for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus antibody (Anti-HCV), anti-HIV antibody, or syphilis antibody.

History of alcohol or drug abuse:

Alcohol: ≥14 units per week; a unit equals 285 mL beer or 100 mL wine. Participants who smoke more than 5 cigarettes/day and cannot stop during the study.

Donation of blood exceeding 400 mL within 1 month prior to the study. Participants enrolled in other drug trials within 3 months before the study. Use of CYP3A4 or P-gp inhibitors/inducers within 28 days prior to the study (e.g., itraconazole, rifampin).

Unwillingness to avoid grapefruit, pomelo, or other food/drinks affecting drug metabolism during the study.

Participants with a history of intestinal surgery affecting drug absorption. Women who are pregnant or lactating or intending to become pregnant. Participants deemed unsuitable by the investigator due to other reasons.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-05-12 (Estimated); Primary Completion 2025-10-12 (Estimated); Study Completion 2026-02-12 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Sudapyridine (WX-081) | From pre-dose Day 1 to Day 7 until post-dose Day 15 to Day 21
  Measurement of the maximum observed plasma concentration of Sudapyridine (WX-081) when administered alone, with itraconazole, with rifampin, and under fasting and fed conditions.
Time to Maximum Plasma Concentration (Tmax) of Sudapyridine (WX-081) | From pre-dose Day 1 to Day 7 until post-dose Day 15 to Day 21
  Measurement of the time to reach the maximum observed plasma concentration of Sudapyridine (WX-081) when administered alone, with itraconazole, with rifampin, and under fasting and fed conditions.
Area Under the Plasma Concentration-Time Curve (AUC0-t and AUC0-∞) of Sudapyridine (WX-081) | From pre-dose Day 1 to Day 7 until post-dose Day 15 to Day 21
  Measurement of the area under the plasma concentration-time curve from time 0 to the last measurable concentration (AUC0-t) and from time 0 extrapolated to infinity (AUC0-∞) of Sudapyridine (WX-081) when administered alone, with itraconazole, with rifampin, and under fasting and fed conditions.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) as Assessed by CTCAE v4.0 | From Day 1 to 7 days post-last dose (up to 35 days, depending on the study part).
  Assessment of treatment-emergent adverse events (TEAEs) using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 to evaluate safety and tolerability.